CLINICAL TRIAL: NCT03273933
Title: DragONE Study: Acquisition and Maintenance of Paediatric Asthma Control: Usual Care vs Innovative Devices
Acronym: DragONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7/2017_B
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 children with DragONE only (Active Comparator)
  Interventions: Device: DragONE
- 10 children with DragONE and SmartOne (Experimental)
  Interventions: Device: DragONE; Device: SmartOne

INTERVENTIONS:
Device: DragONE — The DragONE application for iOS and Android, developed in collaboration with the Institute for Educational Technologies of the National Research Council of Palermo, allow children to daily fill electronically the C-ACT questionnaire and the symptom diary card.
Device: SmartOne — A little portable spirometer connected to DragONE allows daily PEF monitoring.
  Arms: 10 children with DragONE and SmartOne

SUMMARY:
Randomized clinical trial to assess acquisition and maintenance of paediatric asthma control through innovative devices supporting usual care. In the first study arm, a new application (DragONE) for iOS and Android will be only used for patient monitoring. In the second study arm, a small portable device (SmartONE) will also be connected to the DragONE APP, for daily assessment of the peak expiratory flow (PEF). The study duration is 12 weeks. The main outcome of the study is the Childhood Asthma Control Test (C-ACT) score, assessed once every 4 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate persistent asthma
* Uncontrolled symptoms (C-ACT≤ 19)
* Treated for at least 3 months
* FEV1 between 60% and 90% of predicted value

Exclusion Criteria:

* Symptoms of acute respiratory infection
* Immunological or metabolic systemic disease
* Major malformations of the upper airways
* Active smoker

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Acquisition and maintenance of the control status | Once every 4 weeks, for 12 weeks
  mean C-ACT score

SECONDARY OUTCOMES:
Quality of life in asthma children | 12 weeks
  PAQLQ score
Adherence to asthma treatment | 12 weeks
  MARS score
Lung function: FEV1 | 12 weeks
  Forced expiratory volume in the first second
Lung function: FVC | 12 weeks
  Forced vital capacity
Lung function: FEF 25-75 | 12 weeks
  Forced expiratory flow at 25-75%

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM) - National Research Council of Palermo, Palermo, Italy